CLINICAL TRIAL: NCT01189097
Title: Combined Therapy of Methadone and Dextromethrophan: A Novel Strategy for the Treatment of Opioid Dependence
Brief Title: Combined Therapy of Methadone and Dextromethrophan
Acronym: DM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Ru-Band Lu/Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-95-139
Record Dates: First submitted 2010-08-23; First posted 2010-08-26 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2010-08

CONDITIONS: Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dextromethorphan (Experimental)
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan — Subjects who have not used opioid for at least one week before baseline evaluation will take one-week placebo for the wash-out period first and then will be categorized into the opioid free group. The subjects of the opioid using group will be assigned randomly into the following six groups: 1) Methadone + DM 60mg; 2) Methadone + DM 120mg; 3) Methadone + Placebo; 4) Methadone + DM 60mg + motivation and cognitive behavior therapy; 5) Methadone + DM 120mg + motivation and cognitive behavior therapy; 6) Methadone + Placebo + motivation and cognitive behavior therapy. The opioid free group will be 1) DM 30mg; 2) DM 60 mg; 3) Placebo.
Drug: Dextromethorphan — Subjects who have not used opioid for at least one week before baseline evaluation will take one-week placebo for the wash-out period and then randomly assigned into six groups: 1) Methadone + DM 60mg; 2) Methadone + DM 120mg; 3) Methadone + Placebo; 4) Methadone + DM 60mg + motivation and cognitive behavior therapy; 5) Methadone + DM 120mg + motivation and cognitive behavior therapy; 6) Methadone + Placebo + motivation and cognitive behavior therapy. The opioid free group will be 1) DM 30mg; 2) DM 60 mg; 3) Placebo. If the subjects of the opioid free group suffer from relapses and begin to use heroin, they will receive methadone treatment. The dosage of methadone will be increased or decreased maximal 5 mg each time as necessary.

SUMMARY:
The purpose of this study is to determine the pharmacological effects and outcomes of DM therapy with this add-on study.

And to determine the immunological changes between the baseline and the end point of the study.

DETAILED DESCRIPTION:
Opioid dependence is a severe public health problem. Current efforts to taper individuals off opioid medications are limited due to a high relapse rate and lack of efficacy in relieving subjective symptoms. Methadone substitution therapies might decrease the criminal rate and increase the quality of life for individuals with opioid dependence, but the high drop-out rate and continuing use of methadone are major problems in the maintenance of therapy for opioid dependence. Studies in the pathogenesis of opioid dependence and additional behaviors need more focused attention.

Dextromethorphan (DM) is a noncompetitive N-methyl-D-aspartate receptor antagonist that has proven safety record for anti-tussive purpose. Previous studies demonstrated that DM may be useful in decreasing craving in animals (Huang, et al., 2003; Lue et al., 2007) and withdrawal tendencies in human with opioid dependence. In recent studies, DM has been reported to afford neuroprotection against endotoxin-induced dopaminergic neurotoxicity (Li et al. 2005; Liu et al. 2003; Zhang et al. 2004, 2005) which might be related to treatment for additictive behaviors. The purposes of this study are to examine whether DM is able to 1) reduce opioid tolerance and decrease methadone use; 2) reduce withdrawal symptoms; 3) decrease the relapse rate of opioid use, and 4) be an effective treatment for opioid dependence (and addictive behaviors).

This is a double-blinded, placebo-controlled, randomized, and parallel groups clinical research trial study. Subjects with opioid dependence are recruited from two different sources. One group will come from the list of current opioid users and will be required to stay on methadone treatment (opioid using group), and the second group will come from subjects who are forced to discontinue opioid use for more than one week (opioid free group).

In the opioid using group, add-on of DM or placebo treatment will proceed in a double-blind fashion for 12 weeks after completed structured diagnostic interview and adjusted methadone dose. In the opioid free group, subjects will take one-week placebo for the wash-out period first and then will be admitted into a double-blind DM/placebo only for 12 weeks. Both opioid using and opioid free groups will be examined weekly through urine tests for opioid use and will be assessed on a craving scale after the completion of the structured diagnostic interviews. We will measure the treatment response and side effects to clarify the curative effects of DM with the use of the double-blinded DM/placebo therapy design in both the opioid using and opioid free groups. Several psychological examinations, psychosocial questionnaires, tests for immune parameters, electrophysiological studies and genetic markers will be performed in this study. The interim analysis and decording of partial subjects who completed DM/placebo add-on treatment for three months will be performed in the end of first year.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by patient or legal representative.
2. Male or female patient aged ≧18 and ≦65 years.
3. A diagnosis of opioid dependence according to DSM-IV criteria made by a specialist in psychiatry.
4. Patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

1. Women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study.
2. Females who are pregnant or nursing.
3. Patient has received DM or other anti-inflammatory medications within 1 week prior to the first dose of the double-blinded medication.
4. Other major Axis-I DSM-IV diagnosis other than opioid dependence such as multiple substance dependence within 1 year prior to the fist dose of the double-blinded medication.
5. Current evidence of an uncontrolled and/or clinically significant medical condition, e.g., cardiac, hepatic and renal failure that would compromise patient safety or preclude study participation.
6. History of intolerance to methadone or DM.
7. History of sensitivity reaction (e.g., urticaria, angioedema, bronchospasm, severe rhinitis, anaphylactic shock) to DM.
8. Patient has received electroconvulsive therapy (ECT) within 4 weeks prior to the first dose of the double-blinded medication.
9. Increase in total SGOT, SGPT, gamma-GT, BUN and creatinine by more than 3X ULN (upper limit of normal).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-03 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Urinary examination | baseline
  Using urinary examination is aimed to test whether the drug dependence is still using morphine or not.
Urinary examination | week 1
  Using urinary examination is aimed to test whether the drug dependence is still using morphine or not.
Urinary examination | week2
  Using urinary examination is aimed to test whether the drug dependence is still using morphine or not.
Urinary examination | week4
  Using urinary examination is aimed to test whether the drug dependence is still using morphine or not.
Urinary examination | week8
  Using urinary examination is aimed to test whether the drug dependence is still using morphine or not.
Urinary examination | week12
  Using urinary examination is aimed to test whether the drug dependence is still using morphine or not.

SECONDARY OUTCOMES:
cytokines | baseline
cytokines | week1
cytokines | week2
cytokines | week4
cytokines | week8
cytokines | week12

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Band Lu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Ru-Band Lu, Tainan, Taiwan